CLINICAL TRIAL: NCT03225196
Title: Extracellular RNAs in Relation to Cardiometabolic Risk
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999917134; 17-H-N134
Record Dates: First submitted 2017-07-20; First posted 2017-07-21 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Subclinical Atherosclerotic Cardiovascular Disease; Blood Pressure; Obesity
Keywords: Extracellular RNA; MicroRNA; Natural History
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Samples: We seek to measure a 665 exRNAs spanning a variety of classes in plasma from 4095 young to middle-aged adult participants in the Third Generation cohort of the FHS

SUMMARY:
Background:

Extracellular RNAs (exRNAs) send genetic data from cell to cell. This is how they affect the way cells communicate with each other. There are many types of exRNA, and they each serve different roles. But they have also been linked to some diseases. Researchers want to measure exRNAs to see how they relate to certain traits over time. They will use blood samples that were taken as part of the Framingham Heart Study (FHS).

Objectives:

To identify cross-sectional associations of exRNAs with age, sex, and cardiometabolic risk factors.

Eligibility:

People ages 30-70 who had blood taken as part of the FHS Third Generation cohort.

Design:

Researchers will study samples that have already been collected in the FHS. There will be no active participant contact for this project, only use of data that are collected as part of planned follow up from other studies.

As part of the FHS, participants gave blood samples. They gave permission for the blood to be used for research.

The exRNAs from the blood samples will be studied to see how they relate to certain traits. These include age, sex, and body mass index.

The exRNAs will also be studied for their usefulness as biomarkers of risk for subclinical atherosclerotic cardiovascular disease.

No study participants will be contacted for this study....

DETAILED DESCRIPTION:
Extracellular RNAs (exRNAs) impact a wide range of biological processes and function to transfer genetic information between cells. In doing so, exRNAs affect cell-to-cell communications. Recent studies indicate that exRNAs are associated with a variety of diseases. Emerging data from elderly participants in the Framingham Heart Study (FHS) demonstrate that circulating levels of exRNA are correlated with several key traits including age, sex, and body mass index. Much more work is needed to determine the extent to which exRNAs are associated with a variety of clinically relevant traits across the age spectrum. We seek to measure a 665 exRNAs spanning a variety of classes in plasma from 4095 young to middle-aged adult participants in the Third Generation cohort of the FHS and to relate them to age, sex, and cardiometabolic risk factors (BMI, lipids, blood pressure, and fasting glucose) in cross-sectional analyses and to determine the relations of these exRNAs measured at baseline to serial changes in cardiometabolic risk factors during seven years of follow up. We also seek to relate exRNAs to subclinical atherosclerotic cardiovascular disease (ASCVD; assessed via multidetector CT measures of coronary artery calcium), and its progression during seven years of follow up. This grant application will establish an association of exRNAs with clinically relevant traits and diseases and will establish their utility as biomarkers of risk for cardiometabolic disease and subclinical ASCVD. To this end, we propose three aims: 1) To identify associations of exRNAs with age, sex, and cardiometabolic risk factors and subclinical ASCVD at a baseline examination, 2) To identify associations of exRNAs with longitudinal changes in cardiometabolic risk factors and subclinical ASCVD during seven years of follow up, and 3) To explore the genetic regulation of exRNAs via analysis of whole genome sequence data. We demonstrate that we have adequate power to detect associations of exRNAs with cardiometabolic risk factors and subclinical atherosclerosis at baseline and with their longitudinal change during follow up.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:
* FHS Third Generation cohort participants with WGS as part of TOPMed.
* FHS Third Generation cohort participants who attended exam 2 when PaxGene tubes were collected for RNA isolation.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We seek to measure a 665 exRNAs spanning a variety of classes in plasma from 4095 young to middle-aged adult participants in the Third Generation cohort of the FHS
Sampling Method: Non-Probability Sample
Enrollment: 4495 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2020-06-11 (Actual); Study Completion 2020-06-11 (Actual)

PRIMARY OUTCOMES:
subclinical Atherosclerotic disease | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Levy, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- Framingham Heart Study, Framingham, Massachusetts, United States

REFERENCES:
- [Background] Huan T, Rong J, Tanriverdi K, Meng Q, Bhattacharya A, McManus DD, Joehanes R, Assimes TL, McPherson R, Samani NJ, Erdmann J, Schunkert H, Courchesne P, Munson PJ, Johnson AD, O'Donnell CJ, Zhang B, Larson MG, Freedman JE, Levy D, Yang X. Dissecting the roles of microRNAs in coronary heart disease via integrative genomic analyses. Arterioscler Thromb Vasc Biol. 2015 Apr;35(4):1011-21. doi: 10.1161/ATVBAHA.114.305176. Epub 2015 Feb 5. PMID 25657313
- [Background] Tanriverdi K, Kucukural A, Mikhalev E, Tanriverdi SE, Lee R, Ambros VR, Freedman JE. Comparison of RNA isolation and associated methods for extracellular RNA detection by high-throughput quantitative polymerase chain reaction. Anal Biochem. 2016 May 15;501:66-74. doi: 10.1016/j.ab.2016.02.019. Epub 2016 Mar 10. PMID 26969789
- [Background] Yao C, Joehanes R, Johnson AD, Huan T, Esko T, Ying S, Freedman JE, Murabito J, Lunetta KL, Metspalu A, Munson PJ, Levy D. Sex- and age-interacting eQTLs in human complex diseases. Hum Mol Genet. 2014 Apr 1;23(7):1947-56. doi: 10.1093/hmg/ddt582. Epub 2013 Nov 15. PMID 24242183